CLINICAL TRIAL: NCT02458508
Title: Retrospective Evaluation of Prognostic and/or Predictive Profile of Melanocortin Receptor-4 Gene Polymorphisms in Patient With a Diagnosis of Glioblastoma Treated With Upfront Concomitant Radio-chemotherapy or Chemotherapy
Brief Title: Retrospective Evaluation of Melanocortin Receptor 4 Polymorphisms in Patients With GBM Treated With Radiochemotherapy
Acronym: GLIOMELA
Status: Completed | Type: Observational
Sponsor: University of Pisa (Other)
Collaborators: Azienda Ospedaliero, Universitaria Pisana (Other)
Responsible Party: Principal Investigator, Guido Bocci, Asssistant Professor; MD, PhD, University of Pisa
Other Study IDs: University of Pisa
Record Dates: First submitted 2015-05-23; First posted 2015-06-01 (Estimated); Last update posted 2017-10-25 (Actual); Status verified 2017-10

CONDITIONS: Glioblastoma
Keywords: MC4R; chemotherapy; radiotherapy
MeSH Terms: conditions — Glioblastoma

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Biospecimen Retention: Samples With DNA — Blood samples (3 ml) will be collected in EDTA tubes and stored at -80°C from glioblastoma patients
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- GBM patients: patients with diagnosis of glioblastoma treated with concomitant radio-chemotherapy with temozolomide as Stupp protocol will be evaluated for pharmacogenetic evaluation

SUMMARY:
Glioblastoma (GBM) accounts for approximately 50% of all glioma and among these tumors, are the most malignant. The cells of origin of glioma are still undefined, but the most putative target cells include astrocytes, neural stem cells, and oligodendrocyte precursor cells. The current standard of care for patients with newly diagnosed GBM includes temozolomide and radiotherapy . Melanocortins are peptides with well-recognized anti-inflammatory and neuroprotective activity. Of the five known melanocortin receptors (MCRs), only subtype 4 is present in astrocytes and it is expressed predominantly in the brain. No data are currently available on MC4R gene polymorphisms and gliomas or their relationship with radiotherapy or chemotherapy.

Aim. Given the association of MC4R with antiinflammatory activity, neuroprotection, induction of neural stem/progenitor cell proliferation in brain hypoxia, and prevention of astrocyte apoptosis, the aim of this study is to retrospectively evaluate the possible prognostic/predictive role of the MC4R SNPs on GBM therapy.

DETAILED DESCRIPTION:
Glioma is the most frequent malignant primary brain tumor and remains a lethal disease with a dismal prognosis. Glioblastoma (GBM) accounts approximately 50% of all glioma and among these tumors, are the most malignant. GBM are characterized by a higher cellular density and by the ample existence of atypia, mitotic cells, pseudopalisading necrosis and microvascular proliferations. The cells of origin of glioma are still undefined, but the most putative target cells include astrocytes, neural stem cells, and oligodendrocyte precursor cells. Despite therapeutic advances recorded over the last decade, treatment of GBM remains difficult and nowadays no available treatments have a curative attempt. Therefore, the treatment of patients with malignant gliomas still remains palliative. The current standard of care for patients with newly diagnosed GBM was established in 2005 by Stupp et al following the pivotal trial by the European Organisation for the Research and Treatment of Cancer/National Cancer Institute of Canada Clinical Trials Group. The final results of that randomized phase III trial for patients with newly GBM revealed that survival of patients who received temozolomide with radiotherapy for GBM is superior to radiotherapy alone across all clinical prognostic subgroups. On the contrary, the treatment of recurrent GBM is still controversy and continues to be a moving target as new therapeutic principles enrich the standards of care for newly diagnosed disease. After upfront therapy the recurrence rates remain high (≈90%) and the Median overall survival (OS) is 15-18 months in clinical trial populations, and less than 10% of patients are alive at 5 years.

Melanocortins are peptides with well-recognized anti-inflammatory and neuroprotective activity. Of the five known melanocortin receptors (MCRs), only subtype 4 is present in astrocytes. Melanocortin receptor 4 (MC4R) is expressed predominantly in the brain, although it was also detected in adipose tissue, in human skin melanocytes. MC4R has been shown to mediate melanocortin effects on energy homeostasis, reproduction, inflammation, and neuroprotection and, recently, to modulate astrocyte functions. The signaling pathway for MC4R involves G protein-mediated activation of adenylate cyclase and increased cAMP production; in astrocytes it also involves cAMP-protein kinase A (PKA)-cAMP response element binding protein and mitogen-activated protein kinase extracellular signal-regulated kinase -1/2 activation. A recent study showed that melanocyte-stimulating hormone (MSH) induces neurogenesis in the hippocampus of animals after global ischemia and this effect is mediated by MC4R. In an animal model of focal cerebral ischemia, delayed treatment with α-MSH or treatment with Afamelanotide but not with the melanocortin receptor 3 agonist reduced neuron death. This protection correlated with decreased tumor necrosis factor-α and NO production, and decreased expression of pro-apoptotic Bax and caspase-3 activation, and also with increased serum levels of interleukin-10 and Bcl2 expression induced by Afamelanotide. In cerebral ischemia, neuroprotection by Afamelanotide also involves activation of MC4R and Bcl2 upregulation .

Recently, in experimental brain ischemia, treatment with melanocortins acting at melanocortin receptors 4 induces neural stem/progenitor cell proliferation by triggering the canonicalWnt-3A/β-catenin and Shh signaling pathway. Caruso et al. demonstrated that MC4R activation by α-MSH protects astrocytes from apoptosis. Melanocortins prevent astrocyte death by decreasing caspase-3 activity and the expression of Bax and by increasing the expression of Bcl2. As melanocortins increase astrocyte survival, this can contribute to their neuroprotective effects . Moreover, the anti-inflammatory action of α-MSH, an MCR agonist, reduces the secretion of mediators such as cytokines, NO, and prostaglandins and impairs leukocyte activation and infiltration into damaged tissues. Moreover, proliferative effects of α-MSH were reported in 7-day-old cultured astrocytes.

The Single Nucleotide Polymorphisms (SNPs) rs17782313 of the MC4R gene have shown an effect on Body Mass Index (BMI) in different populations; and a direct role in the interaction between Fat Mass and Obesity Associated (FTO) and MC4R gene polymorphisms in breast cancer development has been recently demonstrated. However, no data are currently available on MC4R gene polymorphisms and gliomas or their relationship with radiotherapy/chemotherapy with or without antiangiogenic drugs.

Given the association between MC4R with antiinflammatory activity, neuroprotection, induction of neural stem/progenitor cell proliferation in brain hypoxia, and prevention of astrocyte apoptosis, the aim of this study is to evaluate, retrospectively, the possible prognostic/predictive role of the MC4R SNPs on glioblastoma therapy. Our hypothesis is that these SNPs could have a direct role in the modulation of the therapeutic effects of radiotherapy, chemotherapy and antiangiogenic drugs on glioblastoma and they could influence the prognosis of the disease through their effect on patient's brain.

ELIGIBILITY:
Inclusion Criteria:

* Patients with proven diagnosis of GBM
* Patients suitable for Radio-chemotherapy with temozolomide
* Eastern Cooperative Oncology Group Performance Status 0-2
* Age ≥ 18 years
* Willingness to provide a blood sample for genetic analysis

Exclusion Criteria:

* Patients previously treated with radio or chemotherapy for central nervous system cancer

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with diagnosis of glioblastoma treated with concomitant radio-chemotherapy with temozolomide as Stupp protocol will be evaluated for pharmacogenetic evaluation.
Sampling Method: Non-Probability Sample
Enrollment: 65 (Actual)
Dates: Start 2015-03; Primary Completion 2016-12 (Actual); Study Completion 2017-03 (Actual)

PRIMARY OUTCOMES:
progression-free survival | 12 months
  progression-free survival in GBM patients with different MC4R genotypes and treated with combined radiotherapy and temozolomide

SECONDARY OUTCOMES:
overall survival | 24 months
  overall survival in GBM patients with different MC4R genotypes and treated with combined radiotherapy and temozolomide

CONTACTS AND LOCATIONS:
Overall Officials: Guido Bocci, MD, PhD, Principal Investigator — University of Pisa
Locations (1):
- Division of Radiotherapy, Department Of Oncology, University Hospital of Pisa, Pisa, Italy

REFERENCES:
- [Result] Caruso C, Carniglia L, Durand D, Scimonelli TN, Lasaga M. Astrocytes: new targets of melanocortin 4 receptor actions. J Mol Endocrinol. 2013 Sep 11;51(2):R33-50. doi: 10.1530/JME-13-0064. Print 2013 Oct. PMID 23881919
- [Result] Giuliani D, Minutoli L, Ottani A, Spaccapelo L, Bitto A, Galantucci M, Altavilla D, Squadrito F, Guarini S. Melanocortins as potential therapeutic agents in severe hypoxic conditions. Front Neuroendocrinol. 2012 Apr;33(2):179-93. doi: 10.1016/j.yfrne.2012.04.001. Epub 2012 Apr 17. PMID 22531139
- [Result] Stupp R, Hegi ME, Mason WP, van den Bent MJ, Taphoorn MJ, Janzer RC, Ludwin SK, Allgeier A, Fisher B, Belanger K, Hau P, Brandes AA, Gijtenbeek J, Marosi C, Vecht CJ, Mokhtari K, Wesseling P, Villa S, Eisenhauer E, Gorlia T, Weller M, Lacombe D, Cairncross JG, Mirimanoff RO; European Organisation for Research and Treatment of Cancer Brain Tumour and Radiation Oncology Groups; National Cancer Institute of Canada Clinical Trials Group. Effects of radiotherapy with concomitant and adjuvant temozolomide versus radiotherapy alone on survival in glioblastoma in a randomised phase III study: 5-year analysis of the EORTC-NCIC trial. Lancet Oncol. 2009 May;10(5):459-66. doi: 10.1016/S1470-2045(09)70025-7. Epub 2009 Mar 9. PMID 19269895
- [Result] Preusser M, de Ribaupierre S, Wohrer A, Erridge SC, Hegi M, Weller M, Stupp R. Current concepts and management of glioblastoma. Ann Neurol. 2011 Jul;70(1):9-21. doi: 10.1002/ana.22425. PMID 21786296